CLINICAL TRIAL: NCT02411045
Title: Dress for Success: Can Just Dressing for the Gym Help Going to the Gym?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Harvard University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: 819369-1
Record Dates: First submitted 2015-04-03; First posted 2015-04-08 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-09

CONDITIONS: Healthy
Keywords: Indirect incentives; Exercise more
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- Group 1: Control (Active Comparator): Ask participants to take a picture of themselves
  Interventions: Behavioral: Take and send a selfie
- Group 2: Dress for Success (Experimental): Ask participants to take a picture of themselves while wearing their workout gear
  Interventions: Behavioral: Take and send a selfie; Behavioral: Workout gears
- Group 3: Exercise for Success (Experimental): Ask participants to take a picture of themselves while wearing their workout gear and complete a 30-minute workout
  Interventions: Behavioral: Take and send a selfie; Behavioral: Workout gears; Behavioral: Exercise

INTERVENTIONS:
Behavioral: Take and send a selfie — Direction to take and send a selfie.
Behavioral: Workout gears — Direction to wear workout gears.
  Arms: Group 2: Dress for Success; Group 3: Exercise for Success
Behavioral: Exercise — Direction to complete a 30 minute workout.
  Arms: Group 3: Exercise for Success

SUMMARY:
In this study, the investigators ask the question: can incentivizing smaller, less costly behaviors-like just getting yourself dressed to go to the gym-be more effective (and palatable) than incentivizing the larger goal directly?

DETAILED DESCRIPTION:
To test this hypothesis, the investigators will randomly assign participants to one of three experimental conditions: (1) control, (2) dress for success (low effort), and (2) exercise for success (high effort). The investigators' hypothesis is that incentivizing a low effort, indirect/workout-related behavior (i.e., "dressing for success") will be more effective in motivating workouts than the control, despite a lack of economic incentive for the workout itself. Additionally, the investigators will compare workout levels for groups 2 and 3; if there is no difference between the two groups (or if 2 has higher exercise rates than 3), this would suggest that indirect incentives may be as effective as direct ones.

ELIGIBILITY:
Inclusion Criteria:

* those who opt-in to the recruitment email to all of the investigators' corporate partner's users.

Exclusion Criteria:

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1310 (Actual)
Dates: Start 2015-04; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
number of steps taken | 1-2 weeks before and after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Katherine L. Milkman, Ph.D., Principal Investigator — University of Pennsylvania; Bradford Tuckfield, Principal Investigator — University of Pennsylvania; Katherine Barasz, Principal Investigator — HBS; Leslie K. John, Ph.D., Principal Investigator — HBS
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States